CLINICAL TRIAL: NCT03409458
Title: A Phase 1b/2a Dose Escalation and Confirmation Study of PT-112 in Advanced Solid Tumors in Combination With Avelumab
Brief Title: A Dose Escalation and Confirmation Study of PT-112 in Advanced Solid Tumors in Combination With Avelumab
Acronym: PAVE-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Promontory Therapeutics Inc. (Industry)
Collaborators: Pfizer (Industry); EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-112-103-PAVE-1
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Advanced Solid Tumors; NSCLC; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PT-112 in combination with avelumab (Experimental): PT-112, administered by intravenous infusion avelumab, administered by intravenous infusion
  Patients with all listed conditions are eligible for treatment during the dose escalation phase of the study. Patients with NSCLC are eligible for the dose confirmation phase of the study.
  Interventions: Drug: PT-112; Biological: avelumab

INTERVENTIONS:
Drug: PT-112 — The RP2D of PT-112 when used in combination with avelumab has been determined during dose escalation and is being confirmed in the NSCLC dose confirmation cohort.
  For the NSCLC confirmation cohort, PT-112 will be administered at a dose of 360 mg/m2 on Days 1, 8 and 15.
Biological: avelumab — Avelumab will be administered at a fixed dose of 800 mg on Days 1 and 15.

SUMMARY:
This is a Phase 1/2, open-label, multi-center, non-randomized, dose-escalation study of PT-112 in combination with the anti-PD-L1 antibody, avelumab, in selected advanced solid tumors.

The study is to be conducted in two parts: the Dose Escalation Phase of PT-112 within the combination and the Dose Confirmation Phase in patients with non-small cell lung cancer who will be treated at the RP2D.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, multi-center, non-randomized, dose-escalation study of PT-112 in combination with the anti-PD-L1 antibody, avelumab, in selected advanced solid tumors. The study is to be conducted in two parts: the Dose Escalation Phase and the Dose Confirmation Phase.

Enrollment for dose escalation and dose confirmation is complete.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic or locally advanced, squamous or non-squamous NSCLC (NSCLC). Patients must have received no more than four prior lines of therapy, including a PD-1 / PD-L1-containing therapy and a platinum containing regimen. Patients must have received no more than one taxane containing regimen and no more than one investigational agent;
2. Must provide study-related tumor specimens;
3. ECOG(PS) 0-1;
4. Estimated Life Expectancy > 3 months;
5. Adequate bone marrow (BM), renal, hepatic and metabolic function.

Key Exclusion Criteria:

1. Concurrent cancer treatment with cytoreductive therapy, radiotherapy, cytokine therapy, cytotoxic agents, targeted small molecule therapy or any investigational anticancer small molecule drugs within 2 weeks prior to the start of study treatment (except 5 weeks from last dose of nitrosourea compound) OR treatment with monoclonal antibodies within 4 weeks prior to the start of study treatment;
2. Known symptomatic central nervous system (CNS) metastases requiring steroids.
3. Diagnosis of any other malignancy within 2 years prior to enrollment;
4. Vaccination within 4 weeks of the first dose of study treatment is prohibited except for administration of inactivated vaccines;
5. Current use of immunosuppressive medication at study entry;
6. Active or prior autoimmune disease that might deteriorate with receiving an immunostimulatory agent;
7. Acute or chronic infections requiring systemic therapy;
8. Known history of autoimmune colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis;
9. Known intolerance to checkpoint inhibitor therapy, defined by the occurrence of an AE leading to drug discontinuation;
10. Participation in other studies involving investigational drug(s) within 28 days prior to study entry and/or during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
NSCLC Cohort: Evaluate best overall response rate (ORR) by tumor type according to Immune-Response Criteria (iRECIST) in metastatic or locally advanced, squamous or non-squamous NSCLC. | 24 months

SECONDARY OUTCOMES:
NSCLC Cohort: Confirm the RP2D patients with metastatic or locally advanced, squamous or non-squamous NSCLC | 24 months
NSCLC Cohort: Assess the safety profile of PT-112 in combination with avelumab | 24 months
NSCLC Cohort: Evaluate disease control rate (CR, PR and SD lasting ≥6 months) overall and by tumor type based on iRECIST | 24 months
NSCLC Cohort: Evaluate disease control rate (CR, PR and SD lasting ≥3 months) overall and by tumor type based on iRECIST | 24 months
NSCLC Cohort: Evaluate median duration of response among responding patients | 24 months
NSCLC Cohort: Evaluate median PFS | 24 months
NSCLC Cohort: Evaluate PFS rate at 6 months from start of study drug, based on tumor assessments every 8 weeks based on iRECIST | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Karp, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (5):
  - Arizona, Phoenix, Arizona
  - Colorado, Aurora, Colorado
  - Florida, Jacksonville, Florida
  - Minnesota, Rochester, Minnesota
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Lausanne, Lausanne, Switzerland